CLINICAL TRIAL: NCT04807283
Title: A European Trial Evaluating the Safety and Effectiveness of the Laminar Left Atrial Appendage Closure System in Subjects With Non-Valvular Atrial Fibrillation
Brief Title: Evaluating the Safety and Effectiveness of the Laminar Left Atrial Appendage Closure System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laminar, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CL-0017
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation
Keywords: Left Atrial Appendage Closure
MeSH Terms: conditions — Atrial Fibrillation | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: Left Atrial Appendage Closure

INTERVENTIONS:
Device: Left Atrial Appendage Closure — Closure or occlusion of the left atrial appendage to reduce the risk of thromboembolism in patients with NVAF
  Other Names: Left Atrial Appendage Occlusion

SUMMARY:
The objective of this study is to demonstrate safety and effectiveness using a percutaneous Delivery System of the Laminar Left Atrial Appendage Closure System to treat patients with NVAF to reduce the risk of thromboembolism from the left atrial appendage (LAA).

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject must have a documented history of paroxysmal, persistent or permanent nonvalvular atrial fibrillation (AF).
* 2. Subject must be ≥18 years of age.
* 3. Subject has a calculated CHA2DS2-VASc score of 2 or greater.
* 4. Subject must be clinically stable on warfarin (or other anticoagulant) therapy for a minimum of three months.
* 5. Subject must have at least two International Normalized Ratios (INRs); 2-3, if on Warfarin.
* 6. Subject is eligible for the defined protocol pharmacologic regimen of anticoagulation and antiplatelet therapy.

Exclusion Criteria:

* 1. Subject who requires anticoagulation for a condition other than AF.
* 2. Subject with a New York Heart Association (NYHA) classification equal to IV.
* 3. Subject with a history of or implanted atrial septal defect (ASD) device or patent foramen ovale (PFO) device that would interfere with the investigational device placement.
* 4. Subject with valvular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from device or procedure related serious adverse events | 7 days
Confirmation of functional LAA closure as defined by residual peri-device flow ≤ 5mm per TEE | 45 days

SECONDARY OUTCOMES:
Absence of all-cause mortality, major bleeding, ischemic stroke, or systemic embolism | 45 days and 6 months

CONTACTS AND LOCATIONS:
Locations (4):
- Georgia (2):
  - Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi
  - Tbilisi Heart and Vascular Clinic, Tbilisi
- Paraguay (2):
  - Sanatorio Italiano Hospital, Asunción
  - Hospital de Clinicas San Lorenzo, National University, San Lorenzo

IPD SHARING:
Plan to Share IPD: No